CLINICAL TRIAL: NCT04717791
Title: Low Temperature Controlled Radiofrequency Intranasal Remodeling Treatment of the Nasal Valve Area. A Multicentric Long-term Evaluation
Brief Title: Evaluate the Effectiveness of the Vivaer ARC Stylus for Nasal Breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HNO-Praxis Alte Post (Other)
Collaborators: Aerin Medical (Industry)
Responsible Party: Principal Investigator, Professor Dr. med. Detlef Brehmer, PI Prof. Dr. med. Detlef Brehmer, HNO-Praxis Alte Post
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFNV001
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Nasal Obstruction, Bilateral
Keywords: nasal obstruction; nasal valve stenosis; nasal valve pathology
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Procedure (Other): Subjects will be followed from the Vivaer® treatment date out to 24 months post index procedure.
  Interventions: Device: Vivaer® ARC Stylus

INTERVENTIONS:
Device: Vivaer® ARC Stylus — The Vivaer procedure will be performed in the study clinic using the VivAer Stylus and Aerin Console. The VivAer Stylus is a disposable handheld device capable of delivering low-temperature bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants will have both nasal valves treated in a single study procedure session. Each nostril will be treated at up to 3 positions

SUMMARY:
A Prospective, Multicenter, Non-Randomized Study of the Aerin Medical Vivaer ARC Stylus for Nasal Airway Obstruction

DETAILED DESCRIPTION:
The primary objective of this post-market study is to continue to evaluate the effectiveness of the Vivaer® ARC Stylus for treating the nasal valve area to improve symptoms in those diagnosed with nasal airway obstruction using validated questionaires.

ELIGIBILITY:
Inclusion Criteria:

Eligible subject will meet all the following:

* 1. Age 18 or older 2. Willing and able to provide informed consent 3. Willing and able to comply with the study protocol 4. Seeking treatment for nasal obstruction 5. NOSE score of ≥ 60 at Baseline 6. Nasal valve is a primary or significant contributor to the subject's nasal obstruction as determined by the study investigator (based on clinical presentation, physical examination, nasal endoscopy, etc.) and the subject has a positive response to any of the following temporary measures (based on patient history or office exam):

  * Use of external nasal dilator strips (e.g., Breathe Right Strips)
  * Q-Tip test (manual intranasal lateralization)
  * Use of nasal stents
  * Cottle Maneuver (manual lateral retraction of the cheek)

Exclusion Criteria:

Eligible subjects will NOT meet any of the following:

1. Prior surgical treatment of the nasal valve
2. Rhinoplasty, septoplasty, inferior turbinate reduction or other surgical nasal procedures within the past six months
3. Medical conditions which in the opinion of the treating physician would predispose the subject to poor wound healing or increased surgical risk.
4. Known or suspected to be pregnant or is lactating.
5. Any adjunctive surgical nasal procedure planned on the same day or within 24 months after the Vivaer procedure.
6. Current participation in any study or participation in any study less than 6 weeks before study date 1.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
response rate Nose Score | 3 Months, 6, 12 and 24 months
  The primary efficacy endpoint is the responder rate at 3 months after the procedure for the participants.
  Individual participant success (responder) is defined as at least 1 Nasal Obstruction Symptom Evaluation (NOSE) class improvement or an improvement (decrease) in NOSE score of 20% or more from baseline at the 3-month evaluation.

SECONDARY OUTCOMES:
Efficacy measurement using the change in mean NOSE SCORE | 3 Months, 6, 12 and 24 months
  Efficacy measurement using the change in mean NOSE SCORE from baseline to the 3-month evaluation.
  The Nasal Obstruction Symptom Evaluation (NOSE) scale is a validated disease-specific health status outcomes instrument, used to assess severity of nasal obstruction symptoms. Score ranges from 0 to 100. Higher scores indicate increased symptoms/symptom severity.
Safety Control regarding | 3 Months, 6, 12 and 24 months
  Safety Control regarding the frequency of device-related and procedure-related adverse events.
  All adverse events will be analyzed for all participants. Adverse events will be coded using a custom Aerin Medical dictionary so that adverse events may be categorized for analysis at an appropriate level of detail. Listings will be provided to detail individual events. The number of participants, number of AEs, and the proportion of participants reporting each AE will be summarized. Seriousness and severity of AEs and their relationship to the device and procedure will be summarized. A time course of adverse events will be presented. Any unexpected adverse device experiences or adverse events that occur at an unexpectedly high incidence rate will receive detailed analyses. Narratives will be presented for all deaths, serious adverse events, unexpected adverse device experiences, and participants withdrawn due to an adverse event.

OTHER OUTCOMES:
Adverse events | 3 Months, 6, 12 and 24 months
  Incidence (type and category) of adverse events overall and by follow-up interval.
Nasal Assessment | 3 Months, 6, 12 and 24 months
  The target nasal valve area within each nostril will be visually assessed at baseline and following the treatment procedure at all evaluations. The use of an endoscope for visual assessment is required. Representative still photographs or video of each nostril will be captured at each visit.
Medications | 3 Months, 6, 12 and 24 months
  Self-reported assessment of an increase, no change, or decrease in medications and/or devices being used for treatment of nasal symptoms at each evaluation compared to use prior to the procedure.

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - HNO-Praxis, Lichtenfels, Bavaria
  - HNO-Praxis Alte Post, Göttingen, Niedersachen
  - HNO-ZENTRUM am Kudamm, Berlin

IPD SHARING:
Plan to Share IPD: No